CLINICAL TRIAL: NCT05319717
Title: Rice Bran in Ready-to-use Therapeutic Foods for Microbiota-targeted Treatment of Childhood Malnutrition
Brief Title: Rice Bran-based Supplemental Foods for the Treatment of Childhood Malnutrition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Thrasher Research Fund (Other); Savica, Indonesia (Unknown); Institute of Research for Development, France (Other Government)
Responsible Party: Principal Investigator, Elizabeth P Ryan, Associate Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSU IRB#:1823
Record Dates: First submitted 2022-02-05; First posted 2022-04-08 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Intervention Model Description: Control study arm: Locally produced Ready to use therapeutic food (RUTF)
  Intervention study arm: Locally produced Ready to use therapeutic food plus rice bran (RUTF+RB)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ready-to-use therapeutic food, no rice bran (control/comparator) (Active Comparator): Randomized participants will receive a locally produced ready-to-use therapeutic food to be consumed daily.
  Interventions: Dietary Supplement: Ready-to-use therapeutic food (no rice bran)
- Ready-to-use therapeutic food, with heat stabilized rice bran (Experimental) (Experimental): Randomized participants will receive a locally produced ready-to-use therapeutic food with 5% heat stabilized rice bran to be consumed daily.
  Interventions: Dietary Supplement: Ready-to-use therapeutic food with heat stabilized rice bran

INTERVENTIONS:
Dietary Supplement: Ready-to-use therapeutic food with heat stabilized rice bran — Children assigned to the experimental group will be treated for severe acute malnutrition with a novel ready-to-use therapeutic food that contains 5% heat stabilized rice bran.
  Arms: Ready-to-use therapeutic food, with heat stabilized rice bran (Experimental)
Dietary Supplement: Ready-to-use therapeutic food (no rice bran) — Children assigned to the active comparator group will be treated for severe acute malnutrition with a novel ready-to-use therapeutic food (no rice bran).
  Arms: Ready-to-use therapeutic food, no rice bran (control/comparator)

SUMMARY:
The purpose of this study is to assess the efficacy of treating children with severe acute malnutrition (SAM) with a locally produced ready-to-use therapeutic food (RUTF) with or without rice bran.

DETAILED DESCRIPTION:
Rice bran is a nutrient dense food ingredient with prebiotics and phytochemicals, as well as vitamins, fatty acids, and amino acids. The investigators will determine if the inclusion of rice bran to locally produced RUTFs will improve SAM treatment for children in Indonesia. This will be assessed by standard anthropometric measures and determining the modulation of the malnourished child's gut microbiome and metabolome. The study will also assess rates of relapse in the entire cohort.

This study will yield new information of direct importance and impact to public health nutrition and advance our knowledge and treatment of SAM in Indonesia. Investigation of the gut-microbiota metabolism following consumption of rice bran provided in RUTFs compared to RUTF without rice bran included will provide key mechanistic insights for repairing nutrient absorptive functions in the gut, sustaining gut health in treated children and inform long-term treatment solutions for SAM.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study, with parent(s) signing the informed consent. If the caretaker denies the participation of the child, the child will be enrolled for treatment through the health system, but the information will be not considered for the purpose of the trial.
* Child identified with a weight-for-height z-score WHZ of < -2.5 (SAM children and children with advanced moderate acute malnutrition) and/or mid-upper arm circumference (MUAC) <115 mm) or a child with mild to moderate nutritional edema (regardless of anthropometry).
* Being qualified for outpatient treatment.
* Aged 6-59 months old upon enrolment
* Pass appetite test (taste test) (as stipulated by WHO guidelines on the treatment of SAM). See appetite test document attached.
* Not having consumed RUTF in the last two months

Exclusion Criteria:

* Children detected with severe acute malnutrition younger than 6 months of age will be excluded from the project, as well as any child with a body weight <4.0 kg.
* Children 6-59 months old who, when diagnosed with SAM, have been detected with medical complications, with TB, HIV positive status, one or more signs from the Integrated Management of Childhood Illness (IMCI) guidelines, severe oedema (+++) or who have failed the appetite test (see appetite test document attached).
* Medical complications include: Cough/difficulty in breathing; Diarrhea; Fever; Ear Problems. IMCI signs will be identified according to WHO definition and include not able to drink or breastfeed; vomiting; convulsions; lethargy.
* Participating in another clinical trial
* Any congenital disorder that interferes with normal nutrient intake; chronic conditions including but not exclusively disorders of heart, kidney or liver (children to be screened by a physician).
* SAM with complications requiring hospital treatment. (Upon discharge from hospital, the child will be re-evaluated for inclusion in the study).
* Siblings will not be allowed to participate in the trial

Withdrawal criteria:

* Not consuming the RUTF supplementation at all in >4 days a week in 2 consecutive weeks.
* Not providing samples or completing forms/questionnaires at study visits
* Developing medical complications requiring hospitalization
* Not gaining weight after 1 month of treatment
* Major reactions to intervention

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of the locally produced ready-to-use therapeutic food + heat stabilized rice bran as compared to locally produced ready-to-use therapeutic food alone in the treatment of severe acute malnutrition as determined by child weight. | Baseline, week 4, week 8, and week 16
  This will be assessed by measures of:
  - Weight
Efficacy of the locally produced ready-to-use therapeutic food + heat stabilized rice bran as compared to locally produced ready-to-use therapeutic food alone in the treatment of severe acute malnutrition as determined by mid-upper arm circumference. | Changes between baseline, week 4, week 8, and week 16
  This will be assessed by measures of:
  -Mid-upper arm circumference
Efficacy of the locally produced ready-to-use therapeutic food + heat stabilized rice bran as compared to locally produced ready-to-use therapeutic food alone in the treatment of severe acute malnutrition as determined by morbidity. | Changes between baseline, week 4, week 8, and week 16
  This will be assessed by measures of:
  - Morbidity (diarrhea, fever, vomiting, upper or lower respiratory infection)

SECONDARY OUTCOMES:
Stool microbiota composition | Changes between baseline, week 4, week 8, and week 16
  Determine stool microbiota composition of infants in both arms over time using 16S rRNA sequencing and shotgun metagenomic sequencing.
Dried blood spot metabolite profile | Changes between baseline, week 4, week 8, and week 16
  Dried blood spots will be analyzed for metabolites.
Relapse | Week 16 (end of study)
  Determine the number of participants that experience severe acute malnutrition relapse 4 weeks after the treatment/intervention has ended.
Percent of children recovered | Baseline, week 4, week 8, and week 16
  The number of children recovered in the 4 week treatment period will be determined as well as the time to recovery (days).

CONTACTS AND LOCATIONS:
Overall Officials: Damayanti Soekarjo, PhD, Principal Investigator — Savica, Indonesia
Locations (1):
- Savica, Jember, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
IRB approved study protocol and informed consent forms will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Protocol and informed consent will be shared after enrollment of the first 100 participants
Access Criteria: Sharing access will be made available from the investigative team directly

REFERENCES:
- [Background] Weber AM, Barbazza S, Fauzi MD, Rachmadewi A, Zuhrina R, Putri FK, Campos Ponce M, Hoeven MV, Rimbawan R, Nasution Z, Giriwono PE, Wieringa FT, Soekarjo DD, Ryan EP. Solutions to Enhance Health with Alternative Treatments (SEHAT) protocol: a double-blinded randomised controlled trial for gut microbiota-targeted treatment of severe acute malnutrition using rice bran in ready-to-use therapeutic foods in Indonesia. BMJ Open. 2023 Nov 24;13(11):e076805. doi: 10.1136/bmjopen-2023-076805. PMID 38000818